CLINICAL TRIAL: NCT00003763
Title: A Study to Determine the Ability of Folate Conjugates to Target Folate Receptors in Ovarian Cancer Tumors
Brief Title: Radiolabeled Folic Acid and Imaging to Detect Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocyte (Industry)
Purpose: Diagnostic
Other Study IDs: ENDOCYTE-EC.OV.53.958; CDR0000066889 (Registry Identifier: PDQ (Physician Data Query)); ENDOCYTE-96-286; ENDOCYTE-98-0409
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; ovarian stromal cancer; stage I ovarian germ cell tumor; stage II ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Indium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Procedure: radionuclide imaging
Radiation: indium In 111 folic acid

SUMMARY:
RATIONALE: Diagnostic procedures using the drug radiolabeled folic acid and imaging may be effective in detecting ovarian cancer.

PURPOSE: Diagnostic trial to study the effectiveness of radiolabeled folic acid plus imaging in detecting ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the effectiveness of folic acid conjugated with indium In 111 to diagnose ovarian cancer and locate metastatic disease.

OUTLINE: This is a diagnostic study. Patients receive an injection of folic acid conjugated with indium In 111. The patient then undergoes imaging studies at various time points (e.g., 1, 4, and 24 hours). Patients then undergo exploratory surgery, the results of which are then compared to the imaging studies.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Suspected ovarian cancer OR Recurrence of ovarian cancer Scheduled for exploratory surgery

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3000/mm3 Granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL SGPT and SGOT no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN No acute hepatitis Renal: Creatinine no greater than 1.4 mg/dL BUN no greater than 1.5 times ULN No known or suspected kidney disease Cardiovascular: No history of congestive heart failure No unstable angina No myocardial infarction within 6 months Other: Not pregnant or nursing No septicemia or severe infection No medical condition that would preclude the administration of large fluid volumes over a short period of time

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 3 months since prior cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 months since prior radiotherapy Surgery: See Disease Characteristics Other: At least 2 days since prior folic acid supplements At least 5 days since nonsteroidal antiinflammatory medications

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1997-12-08 (Actual); Primary Completion 2000-05-03 (Actual); Study Completion 2000-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Gershenson, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Washington University - St. Louis, St Louis, Missouri
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No